CLINICAL TRIAL: NCT03744741
Title: HostDx Sepsis in the Diagnosis and Prognosis of Emergency Department Patients With Suspected Infections: a Multicenter Pilot Study
Status: Completed | Type: Observational
Sponsor: Inflammatix (Industry)
Responsible Party: Sponsor
Other Study IDs: OSCCCx-INF-02
Record Dates: First submitted 2018-07-22; First posted 2018-11-16 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Respiratory Tract Infections; Urinary Tract Infections; Skin and Soft Tissue Infections; Intraabdominal Infections; Sepsis
Keywords: Acute Infections; Host response; mRNA; diagnosis; prognosis; procalcitonin; c-reactive protein; molecular respiratory panel; adults
MeSH Terms: conditions — Respiratory Tract Infections; Urinary Tract Infections; Soft Tissue Infections; Intraabdominal Infections; Sepsis; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — PAXgene RNA tubes containing whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: HostDx Sepsis — Blood collection for mRNA analysis, Procalcitonin and CRP determination, molecular analysis of nasopharyngeal swab collection
  Other Names: Procalcitonin; C-reactive protein; Molecular respiratory pathogen panel

SUMMARY:
This study will analyze gene expression data (HostDx Sepsis test) from blood samples collected from participants with suspected infections. The primary endpoint of the study is to prospectively validate the HostDx Sepsis test for infections. As a secondary endpoint the correlation of participant prognosis and gene expression results in the HostDx Sepsis test will be validated. Participants presenting to the emergency departments of enrolling sites with a suspected infection and 1 vital signs OR suspected sepsis and 2 vital sign changes as stated in the protocol are meeting enrollment criteria

DETAILED DESCRIPTION:
Subjects presenting to the emergency department with a suspected acute infection will be eligible. Suspected infections may be of a) respiratory, b) urinary, c) intra-abdominal, or d) skin & soft tissue etiology. Subjects with suspected sepsis of any cause will also be eligible.

Blood sample collections: Clinical study staff or the treating physician will obtain patient consent and collect two PAXgene RNA tubes of whole blood by venipuncture. The blood samples will be stored at room temperature overnight prior to being frozen at -80C for long-term storage. Samples will be shipped to the sponsor for testing using the HostDx Sepsis test. An additional tube of blood obtained via venipuncture and stored for shipment to a centralized testing laboratory, where it will be tested for C-reactive protein and procalcitonin. This will be done for all participants, even if they had these tests ordered locally as SOC.

In participants with suspected respiratory tract infections a nasopharyngeal swab will be collected as intervention and sent to the reference laboratory. The sample will be processed in a respiratory pathogen panel (regardless of whether the participants had or had not provided a nasopharyngeal swab for local testing with a respiratory panel as SOC).

Results obtained from microbiological testing of the following additional samples will be recorded if testing had been performed locally as SOC:

1. Suspected urinary tract infection: Urine sample for culture.
2. Suspected skin & soft tissue infection: Swab from wound or abscess drainage, or other sample, for culture.
3. Suspected intra-abdominal infection or abscesses (e.g. appendicitis, diverticulitis, cholecystitis): Swab, biopsy or other sample types for culture
4. Suspected sepsis of any cause: blood cultures (at least 1 set following local guidelines).
5. Suspected respiratory tract infection: sputum culture and/or throat culture.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 year
2. Suspected Suspected acute infection (respiratory, urinary, abdominal, skin & soft-tissue), and at least one of the symptoms OR, Suspected sepsis of any cause as defined by a blood culture order by the treating physician, and at least two of the symptoms:

   * Heart rate: >90 beats/ minute
   * Temperature: >38 C or <36C
   * Respiratory Rate: >20 breaths / minutes or PaO2 of <60 mmHg or SpO2 <90%
   * Systolic blood pressure: <100 mmHg
   * Altered mental status: Per clinical exam
3. Able to provide informed consent, or consent by legally authorized representative.
4. Subjects in the healthy control group will be eligible if they are i) >18 years of age, ii) able to provide informed consent, iii) in their normal state of health, and iv) do not meet inclusion criteria above

Exclusion criteria:

1. Treatment with systemic antibiotics, antiviral agents, or antifungal agents within the past 7 days prior to the emergency department study visit. Participants will not be excluded for the use topical antibiotics, antiviral agents, or antifungal agents.
2. Prisoners, mentally disabled, or unable or unwilling to give consent.
3. Previously enrolled in the present clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the ED with acute infections or suspected sepsis
Sampling Method: Non-Probability Sample
Enrollment: 585 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Concordance of HostDx Sepsis diagnostic test read-out: likelihood of bacterial infection | 30 days after enrollment
  Percent agreement of HostDx Sepsis bacterial readout with clinical adjudication by physician 30 days after enrollment for the presence of a bacterial infection
Concordance of HostDx Sepsis diagnostic test read-out: likelihood of viral infection | 30 days after enrollment
  Percent agreement of HostDx Sepsis viral readout with clinical adjudication by physician 30 days after enrollment for the presence of a viral infection
Concordance of HostDx Sepsis prognostic read-out (severity) with patient outcome | 30 days after enrollment
  Percent agreement between HostDx Sepsis severity readout and patient outcome, ie mortality, severity of infection, management of patient

CONTACTS AND LOCATIONS:
Locations (7):
- United States (6):
  - Emory University, Atlanta, Georgia
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Baystate Medical Center, Springfield, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Texas Tech University Health Sciences Center El Paso, El Paso, Texas
- Attikon University Hospital, Chaïdári, Greece

IPD SHARING:
Plan to Share IPD: No